CLINICAL TRIAL: NCT00721045
Title: A Phase II Dose-escalation Study to Assess the Feasibility and Safety of Transendocardial Delivery of Three Different Doses of Allogeneic Mesenchymal Precursor Cells (MPCs)in Subjects With Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HF-AB002
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2015-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A1 (Active Comparator): 15 subjects randomized to receive 25 M allogeneic MPCs by transendocardial injection and mapping.
  Interventions: Biological: Mesenchymal Precursor Cells (MPCs)
- A2 (Sham Comparator): 5 subjects randomized to receive standard-of-care treatment with mock mapping and injection procedures.
  Interventions: Procedure: standard-of-care treatment with mock mapping and injection procedures.
- B1 (Active Comparator): 15 subjects randomized to receive 75 M allogeneic MPCs by transendocardial injection and mapping.
  Interventions: Biological: Mesenchymal Precursor Cells (MPCs)
- B2 (Sham Comparator): 5 subjects randomized to receive standard-of-care treatment with mock mapping and injection procedures.
  Interventions: Procedure: standard-of-care treatment with mock mapping and injection procedures.
- C1 (Active Comparator): 15 subjects randomized to receive 150 M allogeneic MPCs by transendocardial injection and mapping.
  Interventions: Biological: Mesenchymal Precursor Cells (MPCs)
- C2 (Sham Comparator): 5 subjects randomized to receive standard-of-care treatment with mock mapping and injection procedures.
  Interventions: Procedure: standard-of-care treatment with mock mapping and injection procedures.

INTERVENTIONS:
Biological: Mesenchymal Precursor Cells (MPCs) — 25 M allogeneic MPCs by transendocardial injection and mapping.
  Other Names: Revascor
  Arms: A1
Biological: Mesenchymal Precursor Cells (MPCs) — 75 M allogeneic MPCs by transendocardial injection and mapping.
  Other Names: Revascor
  Arms: B1
Biological: Mesenchymal Precursor Cells (MPCs) — 150 M allogeneic MPCs by transendocardial injection
  Other Names: Revascor
  Arms: C1
Procedure: standard-of-care treatment with mock mapping and injection procedures. — Mock
  Arms: A2
Procedure: standard-of-care treatment with mock mapping and injection procedures. — Mock
  Arms: B2
Procedure: standard-of-care treatment with mock mapping and injection procedures. — Mock
  Arms: C2

SUMMARY:
This is a dose-ranging clinical study to evaluate the feasibility, safety, and tolerability of 3 different doses of immunoselected, culture expanded, nucleated, allogeneic MPCs in subjects who have cardiomyopathy of both ischemic and idiopathic etiology.

DETAILED DESCRIPTION:
Heart failure subjects recruited will include those who have advanced heart failure NYHA (New York Heart Association) class II to IV and a depressed ejection fraction (EF < 40%). Baseline eligibility testing assessments will be completed within 28 days prior to cell delivery. Efficacy will be explored at 3, 6, and 12 months.

This will be a single-blinded, dose-escalation, cohort study in 60 subjects allocated sequentially to 1 of 3 cohorts A, B, or C. Forty-five subjects will be randomized to receive transendocardial delivery of MPC treatment, and 15 subjects will be randomized to receive standard-of-care treatment without MPC administration. The fifteen subjects randomized to receive standard of care without needle injection will serve as the study's control population and will undergo mock mapping and verbal injection scripts.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA ≥ 2.
2. Age >20 and <80.
3. Cardiomyopathy of ischemic or idiopathic etiology.
4. Subject is not a candidate for either percutaneous intervention or cardiac surgery as determined by both an interventional cardiologist and a cardiac surgeon.
5. LVEF (Left ventricular ejection fraction) < 40% via 2-D Echocardiogram within 28 days of study procedure.
6. On stable maximal, tolerable dosages of heart failure therapies including betablockers,ace inhibitors and/or diuretics with no interruption or change in medical therapy for at least 28 days prior to study enrollment.
7. Left Ventricle wall thickness ≥ 8mm at target site by echo within 28 days of study procedure.
8. If the subject or partner is of childbearing potential, he or she must be willing to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening and for a period of at least 16 weeks after procedure.
9. Female subjects of childbearing potential must have a negative serum pregnancy test at screening.
10. Willing and able to understand, sign, and date the Informed Consent Form (ICF).
11. Must be willing to return for required follow-up visits.
12. Must be able to follow postoperative management program.

Exclusion Criteria:

1. Acute Myocardial Infarction in past 30 days.
2. Discharge of subject's ICD within 28 days of study procedure.
3. Sustained Ventricular Tachycardia as demonstrated by QRS complexes wider than 120 msec, lasting >30 secs, and >100 bpm documented in screening ECG or 24 hour Holter monitoring.
4. Unstable angina.
5. LV thrombus by echocardiogram or angiogram with 28 days prior to and up to the time of cell injection.
6. Aortic stenosis as determined by echocardiography as valve area less than 1 cm2 that prohibits NOGA catheter access to LV.
7. Cardiogenic shock defined as the need for intravenous inotropic support, an intraaortic balloon pump, or mechanical circulatory support at the time of cell injections.
8. Chronic AF or AF at the time of cell injections.
9. Unprotected left main coronary artery disease >50%.
10. Ischemic or hemorrhagic stroke as diagnosed by CT/MRI events within the last 3 months prior to enrollment.
11. Bleeding diathesis disorder such as abnormal coagulation profile precluding performing of mapping/injection procedure.
12. Serum glucose level > 400 mg/dl within 28 days of study procedure.
13. Serum glucose level 300 to 400 mg/dl and presence of urine ketones within 28 days of study procedure.
14. Creatinine level ≥ 2.5 mg/dL within 28 days of study procedure.
15. Hematocrit ≤ 32% within 28 days of study procedure.
16. White Blood Cell count > 12 x 106/mm3 within 28 days of study procedure.
17. Platelet count ≤100 x106/mm3 within 28 days of study procedure.
18. Total bilirubin >3 mg/dL, albumin <2.8 g/dL, aspartate aminotransferase (AST) ≥ 2.5x the upper limit of normal, gamma glutamyltranspeptidase (GGT) ≥ 1.5x the upper limit of normal within 28 days of study procedure.
19. Presence of ≥ 20% anti-HLA antibody titers and/or having antibody specificities to donor HLA antigens.
20. A known hypersensitivity to dimethyl sulfoxide (DMSO), murine and/or bovine products.
21. History of cancer prior to screening (excluding basal cell carcinoma).
22. Acute or chronic infectious disease, including but not limited to human immunodeficiency virus (HIV).
23. Any concurrent disease or condition that, in the opinion of the investigator, would make the subject unsuitable for participation in the study.
24. Treatment and/or an uncompleted follow-up treatment of any investigational. therapy within 6 months before procedure and intent to participate in any other investigational drug or cell therapy study during the 3-year follow-up period of this study.
25. Active participation in other research therapy for cardiovascular repair/regeneration.
26. Prior recipient of stem precursor cell therapy for cardiac repair.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the feasibility and safety of transendocardial injection using mapping Catheter with the Left Ventricular Injection Catheter of 25 M, 75 M, and 150 M allogeneic MPCs in subjects with heart failure. | 3 years

SECONDARY OUTCOMES:
The secondary objectives are to explore functional efficacy for subsequent study design. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD, Principal Investigator — Texas Heart Institute
Locations (6):
- United States (6):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - University of California, San Diego, La Jolla, California
  - Minneapolis Heart Institute 920 East 28th St, Suite 300, Minneapolis, Minnesota
  - UPMC, Pittsburgh, Pennsylvania
  - Texas Heart Institue, Houston, Texas
  - Swedish Heart and Vascular Institute, Seattle, Washington